CLINICAL TRIAL: NCT02576223
Title: Suprascapular Nerve Block as Postoperative Analgesia After Artroscopic Shoulder Surgery - a Randomized, Blinded, Placebo Controlled Study
Brief Title: Suprascapular Nerve Block as Postoperative Analgesia After Artroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kai Henrik Wiborg Lange (Other)
Responsible Party: Sponsor-Investigator, Kai Henrik Wiborg Lange, Head of Research, Hillerod Hospital, Denmark
Organization: Hillerod Hospital, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-15008712; 2015-002391-24 (EudraCT Number)
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pain
Keywords: Peripheral Nerve Blocks
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Sodium Chloride; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine hydrochloride (Active Comparator): Ropivacain 7.5mg/ml, 5 ml injected perineural at the suprascapular nerve.
  Interventions: Drug: Ropivacaine hydrochloride; Drug: PCA-pump
- Isotonic Saline (Placebo Comparator): 0.9% Saline solution, 5 ml injected perineural at the suprascapular nerve.
  Interventions: Drug: Isotonic Saline; Drug: PCA-pump

INTERVENTIONS:
Drug: Ropivacaine hydrochloride — Ropivacaine injected perineural at the suprascapular nerve.
  Other Names: Ropivacaine, Naropin
  Arms: Ropivacaine hydrochloride
Drug: Isotonic Saline — Saline injected perineural at the suprascapular nerve.
  Other Names: Saline
  Arms: Isotonic Saline
Drug: PCA-pump — PCA (Patient controlled analgesia) pump with the following settings:
  Age > 70 years or weight < 60 kg: bolus dose 2,5 mg i.v. morphine, 15 minutes lockout Age < 70 years and weight > 60 kg: bolus dose 5 mg i.v. morphine, 15 minutes lockout Lockout time 15 minutes.
  Other Names: Morphine

SUMMARY:
The purpose of this randomized study is to examine the effect of a selective suprascapular nerve block on post operative pain after arthroscopic shoulder surgery. Half of the subjects will receive a active nerve block with Ropivacain. Half of the subjects will receive a placebo nerve block with saline.

DETAILED DESCRIPTION:
Postoperative pain management after arthroscopic shoulder surgery traditionally includes opioids and/or an interscalene brachial plexus block(IBPB). Opioid consumption often leads to unpleasant side effects including nausea, vomitting and sedation. IBPB offers very efficient pain relief but includes the discomfort of a paralyzed arm. Furthermore this approach often also leads to unilateral paresis of the phrenic nerve causing reduced respiratory capacity. The latter offering discomfort and a potential risk in patients with lung diseases or heavy overweight.

The suprascapular nerve is the most important nerve to the shoulder and a selective block of this nerve could offer a good pain relief without the mentioned side effects.

In this randomized study the investigators wish to examine the pain relieving effect of a selective block of the suprascapular nerve after arthroscopic shoulder surgery.

40 patients are randomized to a block of this nerve with either active drug (Ropivacaine) or placebo (Saline). All patients will get a PCA (Patient Controlled Analgesia) pump for administration of i.v. morphine in doses based on age and weight.

Patient are being monitored for 6 hours. The primary outcome is reduction in VAS at rest from baseline to 30 minutes after nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for arthroscopic shoulder surgery.
* Age ≥ 18.
* ASA class ≤ 3.

Exclusion Criteria:

* Patients with VAS never ≥5 mm during the first hour after arrivel to the post anesthesia care unit.
* Patients unable to cooperate.
* Patients unable to understand or speak danish.
* Allergy towards the used drugs.
* Abuse of alcohol- and/or medicine - investigators assessment.
* Usage of opioids on a daily basis (not including Tramadole).
* Pregnancy (It is obligatory for all fertile women in the study to take a hcg urine test).
* Operations involving the clavicle.
* Operations converted to open surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) score at rest at T½ | Baseline to 30 minutes
  Change in VAS score at rest from baseline to 30 minutes after nerve block (T½).

SECONDARY OUTCOMES:
VAS score during maximum active shoulder abduction from T½ to T6 | ½, 1, 2, 3, 4, 5, 6 hours
  VAS scores measured at 7 timepoints (T½, T1, T2, T3, T4, T5, T6) during maximal active shoulder abduction and calculated as area under the curve (AUC).
VAS score at rest from T½ to T6 | ½, 1, 2, 3, 4, 5, 6 hours
  VAS scores measured at 7 timepoints (T½, T1, T2, T3, T4, T5, T6) at rest and calculated as area under the curve (AUC).
Morphine consumption. | 6 hours
  The total amount of morphine administered via the intravenous PCA pump the first 6 hours after nerve block.
Electromyography at T½ | Baseline to 30 minutes
  Change in activity of the infraspinatus muscle measured with surface electromyography from baseline to T½.
Muscle strength at T½ | Baseline to 30 minutes
  Change in strength of the supraspinatus (abduction of the shoulder) and the infraspinatus muscle (external rotation of the shoulder) measured with a handheld dynamometer from baseline to T½.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Steen-Hansen, Principal Investigator — Nordsjaellands Hospital
Locations (2):
- Denmark (2):
  - Nordsjællands Hospital, Hillerød
  - Holbæk Sygehus, Holbæk